CLINICAL TRIAL: NCT02130219
Title: Scientific Research and Development of Innovative Evidence Based Non-invasive Brain Diagnostic and Monitoring Solutions for Neurological and Traumatic Brain Injury Patients
Brief Title: Clinical Value of Noninvasive Intracranial Pressure Measurement
Acronym: Braincare
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Principal Investigator, Kestutis Petrikonis, M.D., PhD, Associated professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CH-3-SMM-01/06; BE-2-26 (Other Grant/Funding Number: Regional bioethics commitee)
Record Dates: First submitted 2014-03-20; First posted 2014-05-05 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-03

CONDITIONS: Intracranial Hypertension
Keywords: ICP, intracranial hypertension, Vittamed 205
MeSH Terms: conditions — Intracranial Hypertension | interventions — Spinal Puncture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chronic daily headache group (Experimental): Patients with chronic daily headache with suspicion of intracranial hypertension selected. Selection based on clinical symptoms (headache description, leading symptoms)and para-clinical pathological findings (optical nerve papilla edema). Not enough evidence to diagnose any other headache type. Simultaneous CSF pressure measurements and non-invasive ICP measurement will be performed.
  Interventions: non-invasive intracranial pressure measurement; lumbar puncture and cerebrospinal fluid pressure measurement; brain MRI/CT.
  Interventions: Device: Non-invasive intracranial pressure measurement; Device: Brain MRI/CT; Procedure: Lumbar puncture and cerebrospinal fluid pressure measurement
- Multiple sclerosis group (Experimental): Multiple sclerosis (MS) group patients selected based on clinical symptoms and brain MRI changes typical for the disease. Diagnosis based on McDonalds criteria. CSF test for oligoclonal bands required as supporting diagnostic criteria. Patients selected with disease relapse symptoms. Simultaneous noninvasive ICP and CSF pressure measured.
  Interventions: non-invasive intracranial pressure measurement; lumbar puncture and cerebrospinal fluid pressure measurement; brain MRI/CT
  Interventions: Device: Non-invasive intracranial pressure measurement; Device: Brain MRI/CT; Procedure: Lumbar puncture and cerebrospinal fluid pressure measurement
- Stroke group (Experimental): Patients selected for this group have stroke/intracranial hemorrhage that might be complicated with intracranial hypertension. Stroke/intracranial hemorrhage diagnosed based on clinical findings and changes on brain CT/MRI. Patients with stroke less than 33% of middle cerebral artery territory included. Patients with intracranial hemorrhage 20-40 ml volume included. Patients unable to cooperate or sign informed consent excluded.
  Bilateral non-invasive ICP measurements performed. Results compared with brain MRI/CT lesion volume, mid-line shift.
  Interventions: non-invasive intracranial pressure measurement; brain MRI/CT
  Interventions: Device: Non-invasive intracranial pressure measurement; Device: Brain MRI/CT
- Normal pressure hydrocephalus group (Experimental): Patients meeting normal pressure hydrocephalus diagnosis criteria selected to compare invasive CSF pressure versus non-invasive ICP.
  Interventions: non-invasive intracranial pressure measurement; lumbar puncture and cerebrospinal fluid pressure measurement; brain MRI/CT
  Interventions: Device: Non-invasive intracranial pressure measurement; Device: Brain MRI/CT; Procedure: Lumbar puncture and cerebrospinal fluid pressure measurement

INTERVENTIONS:
Device: Non-invasive intracranial pressure measurement — The noninvasive ICP measurement device Vittamed 205 aICP meter used in this study has been developed in Lithuania. The method is based on two-depth transcranial Doppler technique for simultaneously measuring flow velocity pulsatilities in the intracranial and extracranial segments of the ophthalmic artery (OA). These measurements are made while applying a series of small pressure steps to the tissues surrounding the eye-ball. The intracranial segment of the OA is compressed by ICP and the extracranial segment of the OA is compressed by the externally applied pressure Pe. Blood flow pulsatility parameters in both of these OA segments are monitored.Pulsatilities are approximately the same when Pe = ICP. Two-depth TCD device is used as an indicator of the pressure balance point.
  Other Names: Non-invasive aICP meter Vittamed 205
Device: Brain MRI/CT — 1.5 T MRI using T1 and T2 regimes, brain MRI angiography, performed for selected patients to analyze anatomical features of ophthalmic artery and optical nerves sheath diameter.
  Brain CT performed to evaluate hemorrhage and stroke volume.
Procedure: Lumbar puncture and cerebrospinal fluid pressure measurement — Lumbar puncture performed in lateral decubitus position while knees and head flexed. After local antiseptics and anesthesia puncture in lumbar 3/4 or 4/5 intervertebral space performed. As CSF appears legs and head are relaxed and slightly straightened. Spinal manometer graded 0-40 cm H₂O with stopcock connected to the needle. CSF pressure monitored for 10 minutes and recorded. CSF collected for diagnostic test. Spinal needle Number 22 and Rocket Spinal Manometer Set (No. R55990) used for this study.
  Other Names: CSF pressure measurement
  Arms: Chronic daily headache group; Multiple sclerosis group; Normal pressure hydrocephalus group

SUMMARY:
The aim of the study is to evaluate accuracy and precision of non-invasive intracranial pressure measurement device (Vittamed 205) for selected patients compared with cerebrospinal fluid pressure measured during lumbar puncture

DETAILED DESCRIPTION:
Non-invasive intracranial pressure (ICP) measurements with Vittamed 205 aICP meter will be compared to simultaneous cerebrospinal fluid (CSF) pressure measurements during lumbar puncture. Measures of pressure in mmHg will be compared. These measurements will be compared in chronic daily headache, normal pressure hydrocephalus and multiple sclerosis patients groups. For stroke patients noninvasive measurements will be compared with cerebral lesion in brain MRI/CT.

ELIGIBILITY:
Inclusion Criteria:

* Chronic daily headache with suspected idiopathic intracranial hypertension
* Diagnosed of suspected multiple sclerosis (MS)
* Intracranial hemorrhage/ stroke

Exclusion Criteria:

* Patient not able to understand information about the trial
* Uncooperative patient
* Intracranial hemorrhage volume <20 or >40ml
* Stroke area larger than 1/3 of the middle cerebral artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the results of noninvasive intracranial pressure measurement (with Vittamed 205 aICP meter) within clinically acceptable 4 mm Hg difference from invasively measured CSF pressure. | Simultaneous noninvasive ICP and CSF pressure measurements. All measurements will be collected within 20 months until 31 December 2014.
  Brain MRI/CT data will be used to compare ocular nerve sheath diameter (in mm) and stroke/ intracerebral hemorrhage volume (in cubic cm) with CSF pressure and non-invasive ICP.

CONTACTS AND LOCATIONS:
Overall Officials: Kestutis Petrikonis, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania

REFERENCES:
- [Background] Ragauskas A, Bartusis L, Piper I, Zakelis R, Matijosaitis V, Petrikonis K, Rastenyte D. Improved diagnostic value of a TCD-based non-invasive ICP measurement method compared with the sonographic ONSD method for detecting elevated intracranial pressure. Neurol Res. 2014 Jul;36(7):607-14. doi: 10.1179/1743132813Y.0000000308. Epub 2014 Jan 12. PMID 24620972
- [Background] Ragauskas A, Matijosaitis V, Zakelis R, Petrikonis K, Rastenyte D, Piper I, Daubaris G. Clinical assessment of noninvasive intracranial pressure absolute value measurement method. Neurology. 2012 May 22;78(21):1684-91. doi: 10.1212/WNL.0b013e3182574f50. Epub 2012 May 9. PMID 22573638